CLINICAL TRIAL: NCT02779192
Title: A Phase 2b, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety and Efficacy of SPI-1005 to Prevent Acute Noise Induced Hearing Loss (PANIHL)
Brief Title: A Phase 2b Study of SPI-1005 to Prevent Acute Noise Induced Hearing Loss
Acronym: PANIHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-1005-203
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Noise Induced Hearing Loss
Keywords: Acute Noise Induced Hearing Loss; Prevent Acute Noise Induced Hearing Loss
MeSH Terms: conditions — Hearing Loss, Noise-Induced | interventions — ebselen; Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SPI-1005 200 mg (Active Comparator): 200 mg SPI-1005, capsule, bid, po, x7d
  Interventions: Drug: SPI-1005 200mg
- SPI-1005 400 mg (Active Comparator): 400 mg SPI-1005, capsule, bid, po, x7d
  Interventions: Drug: SPI-1005 400mg
- Placebo (Placebo Comparator): 0 mg SPI-1005, capsule, bid, po, x7d
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPI-1005 200mg — Oral SPI-1005 capsules, 200 mg ebselen, twice daily, 7 days
  Other Names: Low Dose
  Arms: SPI-1005 200 mg
Drug: SPI-1005 400mg — Oral SPI-1005 capsules, 400 mg ebselen, twice daily, 7 days
  Other Names: High Dose
  Arms: SPI-1005 400 mg
Drug: Placebo — Oral SPI-1005 capsules, 0 mg ebselen, twice daily, 7 days
  Other Names: Control
  Arms: Placebo

SUMMARY:
SPI-1005 is a novel oral drug that contains a glutathione peroxidase mimetic (ebselen) that will be tested in subjects with a history of NIHL at risk for additional NIHL. The goal of this multi-center Phase 2b study is to determine whether SPI-1005 is effective in reducing an acute NIHL in this affected population. In this Phase 2b study subjects with prior NIHL will be enrolled and exposed to a calibrated sound challenge (CSC) that induces a slight acute NIHL.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, safety and efficacy study of oral SPI-1005 in adults with Noise Induced Hearing Loss (NIHL). All recruited subjects will have their severity of NIHL determined before the start of SPI-1005 treatment using various hearing tests. Subjects will be enrolled and randomized to either placebo or SPI-1005. Subjects will be dosed with either placebo or SPI-1005 for 7 days, beginning 1 day before an acute NIHL. Subjects will have hearing tests performed before and immediately after a calibrated sound challenge (CSC). Follow-up hearing tests will be performed post-CSC.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients, 18-50 years of age
* History of either recreational and/or occupational exposure to noise
* Voluntarily consent to participate in the study
* Females of childbearing potential should be using and committed to continue using one of the following acceptable birth control methods: Sexual abstinence (inactivity) for 14 days prior to screening through study completion; or intra-uterine device in place for at least 3 months prior to study through study completion; or barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through study completion; or stable hormonal contraceptive for at least 3 months prior to study through study completion; or surgical sterilization (vasectomy) of partner at least 6 months prior to study.
* Females of non-childbearing potential should be surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to study, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be at least 3 years since last menses.

Exclusion Criteria:

* Current use or within 60 days prior to study of excluded ototoxic medications
* History of autoimmune inner ear disease
* History of middle ear or inner ear surgery
* Current conductive hearing loss or middle ear effusion
* Significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, or psychiatric disease
* History of hypersensitivity or idiosyncratic reaction to compounds related to ebselen
* Current use or within 30 days prior to study of drugs or substances known to be strong inhibitors or inducers of cytochrome P450 enzymes
* Participation in another investigational drug or device study within 90 days prior to study enrollment
* Female patients who are pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in the Incidence of a Significant Threshold Shift | Within 1 day
  Post Controlled Sound Challenge pure tone audiometry will be compared with baseline

SECONDARY OUTCOMES:
Improvement in word recognition score | Within 1 day
  Post Controlled Sound Challenge Words in Noise Test score will be compared with baseline

OTHER OUTCOMES:
Adverse events | Within 7 days
  Adverse events due to study drug will be compared with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kil, MD, Study Chair — SOUND PHARMACEUTICALS, INC.
Locations (5):
- United States (5):
  - University of Miami, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - MUSC, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - Sound Pharmaceuticals, Inc., Seattle, Washington

IPD SHARING:
Plan to Share IPD: No